CLINICAL TRIAL: NCT00083317
Title: The Role of the Prefrontal Cortex in Economic Decision-Making in Reciprocal Trust Games Using Functional Hyperscanning Neuroimaging
Brief Title: Role of the Brain in Making Economic Decisions
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040192; 04-N-0192
Record Dates: First submitted 2004-05-19; First posted 2004-05-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-01-04

CONDITIONS: Healthy
Keywords: PFC; Competition; Bargaining Games; Hyper-Brain Scanning; fMRI; Healthy Volunteer; HV

SUMMARY:
This study will identify which areas of the brain mediate the interaction between people involved in economic decision-making.

Healthy, right-handed native English speakers between 21 and 55 years of age may be eligible for this study. Candidates are screened with a telephone interview, a questionnaire to determine handedness, and a neurological examination if one has not been performed within the last year by an NIH physician.

Participants bargain for money by playing two-person trust games, while undergoing functional magnetic resonance imaging (fMRI). MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the procedure, the subject lies on a stable that can slide in and out of the scanner, wearing earplugs to muffle loud knocking sounds that occur with electrical switching of the magnetic fields. Functional MRI involves taking MRI scans while the subject performs a task-this to learn about how the brain regions are involved in performing the task. For this test, the subject plays or watches two-person games involving trust. The game may be played against a stranger or a friend. The winner receives a cash payoff.

The subject performs one of the following two tasks during MRI scanning:

* Playing the trust games and indicating as quickly as possible by pressing a right or left button whether he or she wants to stop or continue playing, or
* Observing games that others have played and predicting as quickly as possible by pressing a right or left button whether the players wanted to stop or continue the games.

The test takes about 90 minutes. After the scan, participants complete written questionnaires about their experience in the scanner and their views on issues related to participating in competitive games.

...

DETAILED DESCRIPTION:
Objective. The purpose of the protocol is to identify the brain regions mediating the social cooperation involved in economic decision-making, including whether negative mood and perceived interpersonal similarity affect behavior or brain regions utilized.

Study Population. Healthy, normal adult volunteers will play and observe two-person reciprocal trust games during functional neuroimaging against either real people or computers masquerading as real people.

Design. A between/within-subject, rapid event-related fMRI design will be employed for two series of experiments. In the first experiment, two persons-each in a separate MRI scanner-will interact with one another playing two-person reciprocal trust games while their brains are simultaneously scanned. In the second experiment, a third person will later observe the played games while in a scanner, trying to predict the decisions of the two other players in the first experiment. In the third experiment, a sad mood will be induced in half of the participants to examine if it affects levels of cooperative behavior and patterns of brain activation in the two types of trust games described above.

Four additional series of experiments will employ between/within subject designs in which subjects are scanned alone, but under the deception that they are playing simultaneously with another subject.

Outcome Measures. The data collected will consist of behavioral measures of cognitive performance, self- and other-mental representation, trusting and trustworthy behavior, corresponding fMRI images, personality scales, ratings of relationship and status, and types of strategy used. The results gained from this protocol will be of value in identifying a set of neural regions mediating dynamic social interaction between people engaged in economic decision-making.

ELIGIBILITY:
* INCLUSION CRITERIA:

In all the studies, subjects will consist of healthy, native English-speaking, right-handed volunteers, as measured by the Edinburgh Handedness Inventory (Oldfield, 1971). Subjects will range in age from 21 to 55 years old and they will be included regardless of race.

EXCLUSION CRITERIA:

Non-native English speakers and non-right handers will be excluded as mentioned above, as will non-neurologically normal volunteers. Subjects younger than 21 and older than 55 will be excluded. A urine pregnancy test will be employed with all women of childbearing age. The results must be negative in order to proceed with the MRI.

Participants with any of the following: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body, e.g. metal shavings; permanent eyeliner; insulin pump; or irremovable body piercing will be excluded from the study due to the possible dangerous effects of the magnet upon metal objects in the body. Participants taking central nervous system active medications will be excluded.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2004-05-15; Study Completion 2012-01-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bell AJ, Sejnowski TJ. An information-maximization approach to blind separation and blind deconvolution. Neural Comput. 1995 Nov;7(6):1129-59. doi: 10.1162/neco.1995.7.6.1129. PMID 7584893
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.
- [Background] Belliveau JW, Rosen BR, Kantor HL, Rzedzian RR, Kennedy DN, McKinstry RC, Vevea JM, Cohen MS, Pykett IL, Brady TJ. Functional cerebral imaging by susceptibility-contrast NMR. Magn Reson Med. 1990 Jun;14(3):538-46. doi: 10.1002/mrm.1910140311. PMID 2355835